CLINICAL TRIAL: NCT04207346
Title: Transcranial Magnetic Stimulation to Improve Functioning in Veterans With PTSD
Acronym: rTMS for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2905-R
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: PTSD
Keywords: Transcranial Magnetic Stimulation; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study: procedure vs. sham procedure
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS (Experimental): transcranial magnetic stimulation delivered to the right dorsolateral prefrontal cortex at 1 Hz
  Interventions: Device: TMS 1 hz
- Sham (Sham Comparator): sham transcranial magnetic stimulation delivered to the right dorsolateral prefrontal cortex
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: TMS 1 hz — High-performance magnetic stimulator designed for clinical use or use in clinical trials. This specific device has a coil designed with one side that delivers active treatment and the other side that delivers sham (no stimulation) treatment. The sham side is externally identical to the active side, but internally it has a shield that prevents any magnetic energy from interacting with the patient. This arm will use the active side.
  Other Names: MagPro R30 TMS device produced by MagVenture
  Arms: TMS
Device: Sham TMS — High-performance magnetic stimulator designed for clinical use or use in clinical trials. This specific device has a coil designed with one side that delivers active treatment and the other side that delivers sham (no stimulation) treatment. The sham side is externally identical to the active side, but internally it has a shield that prevents any magnetic energy from interacting with the patient. This arm will use the sham side.
  Other Names: MagPro R30 TMS device produced by MagVenture
  Arms: Sham

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is a common and serious condition affecting many Veterans. There are effective treatments for PTSD, but additional treatments are needed in order to better serve Veterans suffering from PTSD. Transcranial magnetic stimulation is one such promising treatment. It involves use of powerful magnet to stimulate the specific brain regions in Veterans with PTSD. Transcranial magnetic stimulation has been shown effective in treating depression, but currently it is unclear if it is an effective treatment for PTSD. This is a randomized clinical trial enrolling 91 Veterans with PTSD comparing the effectiveness of transcranial magnetic stimulation treatment and sham transcranial magnetic stimulation in treating PTSD. The hypothesis is that those who receive transcranial magnetic stimulation will experience improved functioning.

DETAILED DESCRIPTION:
Background Posttraumatic Stress Disorder (PTSD) is an often chronic and disabling condition prevalent in the Veteran population. While there is sufficient evidence to demonstrate the effectiveness of medications and psychotherapy for improving PTSD symptoms, there has been limited study of functioning as an outcome, and the role of other treatments such as somatic therapies. One promising but understudied somatic treatment for PTSD is repetitive transcranial magnetic stimulation (TMS). The characteristics of TMS treatment are different than those of existing treatments and may provide alternative treatment to Veterans who do not respond to medications and psychotherapy. Further, it is possible that TMS may have a greater effect on functioning and lead to higher rates of recovery compared with medications or psychotherapy.

Objective To determine whether Veteran participants with PTSD who receive TMS delivered to the right dorsolateral prefrontal cortex at 1 Hz have greater improvements in: PTSD symptoms, functioning, and depressive symptoms than Veterans receiving sham treatments at treatment completion and at 3 and 6 months after treatment completion.

Method 91 Veterans with PTSD will be randomly assigned to receive low frequency TMS or sham TMS. All TMS will be applied to the right dorsolateral prefrontal cortex. PTSD symptoms, functional outcomes, and depressive symptoms will be measured for all participants at treatment completion, 3 months, and 6 months after completion.

Hypothesis Veterans with PTSD receiving TMS will have greater improvements in PTSD symptoms, functioning, and depressive symptoms at treatment completion and at three and six months after treatment completion compared to Veterans receiving sham TMS.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 19 and 70
2. Moderate to severe PTSD as determined by the CAPS within 7 days of randomization.
3. Agree to have CAPS audio-recorded.
4. Ability to obtain a Motor Threshold using the TMS device during screening.
5. Patient eligible for VA healthcare.
6. If female with childbearing potential, use of acceptable method of birth control (i.e., use of contraceptives, abstinence).
7. Able to read, understand, and sign the informed consent document.

Exclusion Criteria:

1. Pregnant or lactating woman.
2. Current use of clozapine (any dose) or bupropion (more than 300mg per day).
3. Cardiac pacemaker or implantable defibrillator.
4. Presence of any metal object in the head, including cochlear implants, but excluding dental work in the mouth.
5. Significant central nervous system disorder (stroke, brain mass, epilepsy).
6. Seizure in past one year.
7. Current psychosis or mania.
8. Prior use of TMS.
9. Significant suicidal ideation.
10. Unstable medical conditions.
11. Current alcohol or substance use disorder (except nicotine) that interferes with the patient's ability to participate.
12. CPT or PE for PTSD in the past 2 months.
13. Changes in Fluoxetine, Paroxetine, Sertraline, or Venlafaxine in the past 2 months.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
CAPS | Baseline
  The Clinician-administered scale of PTSD symptoms (CAPS) queries the frequency and intensity of symptoms of PTSD. The score ranges from 0-80 with a higher score indicating worse symptoms. It is considered the gold standard for diagnosis and symptoms assessment in PTSD clinical studies.
WHODAS | Baseline
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) is a 36 item self-report instrument that assesses disability and function across six domains: communicating, getting around, self-care, getting along with people, life activities, and participation in society. The WHODAS has been used as an outcome of function and disability across many disorders and is commonly used in mental health treatment trials. The total score ranges from 0-100 with a higher score indicating worse functioning.
QIDS SR-16 | Baseline
  The Quick Inventory of Depressive Symptomatology (QIDS SR-16) is a 16-item self-report measure of depression. The QIDS SR-16 includes nine domains that relate to the nine primary symptoms of major depressive disorder in the DSM-IV. The score ranges from 0-27 with a higher score indicating worse depression.
CAPS | 2 weeks
  The Clinician-administered scale of PTSD symptoms (CAPS) queries the frequency and intensity of symptoms of PTSD. The score ranges from 0-80 with a higher score indicating worse symptoms. It is considered the gold standard for diagnosis and symptoms assessment in PTSD clinical studies.
CAPS | 3 months
  The Clinician-administered scale of PTSD symptoms (CAPS) queries the frequency and intensity of symptoms of PTSD. The score ranges from 0-80 with a higher score indicating worse symptoms. It is considered the gold standard for diagnosis and symptoms assessment in PTSD clinical studies.
CAPS | 6 months
  The Clinician-administered scale of PTSD symptoms (CAPS) queries the frequency and intensity of symptoms of PTSD. The score ranges from 0-80 with a higher score indicating worse symptoms. It is considered the gold standard for diagnosis and symptoms assessment in PTSD clinical studies.
WHODAS | 2 weeks
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) is a 36 item self-report instrument that assesses disability and function across six domains: communicating, getting around, self-care, getting along with people, life activities, and participation in society. The WHODAS has been used as an outcome of function and disability across many disorders and is commonly used in mental health treatment trials. The total score ranges from 0-100 with a higher score indicating worse functioning.
WHODAS | 3 months
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) is a 36 item self-report instrument that assesses disability and function across six domains: communicating, getting around, self-care, getting along with people, life activities, and participation in society. The WHODAS has been used as an outcome of function and disability across many disorders and is commonly used in mental health treatment trials. The total score ranges from 0-100 with a higher score indicating worse functioning.
WHODAS | 6 months
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) is a 36 item self-report instrument that assesses disability and function across six domains: communicating, getting around, self-care, getting along with people, life activities, and participation in society. The WHODAS has been used as an outcome of function and disability across many disorders and is commonly used in mental health treatment trials. The total score ranges from 0-100 with a higher score indicating worse functioning.
QIDS SR-16 | 2 weeks
  The Quick Inventory of Depressive Symptomatology (QIDS SR-16) is a 16-item self-report measure of depression. The QIDS SR-16 includes nine domains that relate to the nine primary symptoms of major depressive disorder in the DSM-IV. The score ranges from 0-27 with a higher score indicating worse depression.
QIDS SR-16 | 3 months
  The Quick Inventory of Depressive Symptomatology (QIDS SR-16) is a 16-item self-report measure of depression. The QIDS SR-16 includes nine domains that relate to the nine primary symptoms of major depressive disorder in the DSM-IV. The score ranges from 0-27 with a higher score indicating worse depression.
QIDS SR-16 | 6 months
  The Quick Inventory of Depressive Symptomatology (QIDS SR-16) is a 16-item self-report measure of depression. The QIDS SR-16 includes nine domains that relate to the nine primary symptoms of major depressive disorder in the DSM-IV. The score ranges from 0-27 with a higher score indicating worse depression.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley V Watts, MD MPH, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (1):
- White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No